CLINICAL TRIAL: NCT07323641
Title: A Phase II Trial of Telisotuzumab Vedotin With Osimertinib for EGFR Mutated NSCLC With c-MET Overexpression That is Progressing on Osimertinib
Brief Title: Telisotuzumab Vedotin and Osimertinib for the Treatment of Progressive, Incurable, Non Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-2145; NCI-2025-09155 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2026-01-06; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; osimertinib; telisotuzumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (telisotuzumab vedotin and osimertinib) (Experimental): Patients receive telisotuzumab vedotin IV on days 1 and 15 of cycles 1-3 and on day 1 of subsequent cycles. Patients also receive osimertinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, brain MRI, if needed, and blood sample collection throughout the study. Patients also optionally undergo tumor biopsy during follow-up.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Osimertinib; Other: Survey Administration; Biological: Telisotuzumab Vedotin

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Osimertinib — Given PO
  Other Names: AZD 9291; AZD-9291; AZD9291; Mereletinib
Other: Survey Administration — Ancillary studies
Biological: Telisotuzumab Vedotin — Given IV
  Other Names: ABBV 399; ABBV-399; ABT 399; ABT-399; ABT-700-VCMMAE; Emrelis; Telisotuzumab Vedotin-tllv

SUMMARY:
This phase II trial tests how well telisotuzumab vedotin and osimertinib works for the treatment of non small cell lung cancer that is growing, spreading, or getting worse (progressive) and for which no treatment is currently available (incurable). Telisotuzumab vedotin is a monoclonal antibody, called telisotuzumab, linked to a toxic agent, called vedotin. Telisotuzumab is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of tumor cells, known as c-Met receptors, and delivers vedotin to kill them. Osimertinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving telisotuzumab vedotin and osimertinib may be effective for treating progressive, incurable non small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Objective response rate (ORR) as defined as complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.

II. Progression free survival (PFS) as defined by time from treatment initiation to disease progression per RECIST 1.1 criteria or death.

SECONDARY OBJECTIVES:

I. Duration of response (DOR), time to response (TTR) and overall survival (OS).

II. Assess the safety and tolerability of induction and maintenance schedule of telisotuzumab vedotin when given with osimertinib in all evaluable patients who received at least one dose of study regimen.

EXPLORATORY OBJECTIVES:

I. Assess potential biomarkers associated with response from liquid biopsies and archival or fresh tissue biopsy.

Ia. Correlate tissue biomarkers such as MET expression level by immunohistochemistry and ribonucleic acid (RNA) expression with response; Ib. Where an archival specimen is available from prior to treatment with an EGFR tyrosine kinase inhibitor (TKI) and can be compared to a more recent specimen, the dynamics and predictive value of c-MET overexpression will be evaluated.

II. Assess participant-reported outcomes on quality of life using Functional Assessment of Cancer Therapy-Lung Cancer Subscale (FACT-LCS) questionnaire.

OUTLINE:

Patients receive telisotuzumab vedotin intravenously (IV) on days 1 and 15 of cycles 1-3 and on day 1 of subsequent cycles. Patients also receive osimertinib orally (PO) daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) scan, brain magnetic resonance imaging (MRI), if needed, and blood sample collection throughout the study. Patients also optionally undergo tumor biopsy during follow-up.

After completion of study treatment, patients are followed up at 30 days and every 6 weeks or 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age and willing and able to provide informed consent
* Cytologically or histologically confirmed non small cell lung cancer (NSCLC), which is incurable with an activating and sensitizing EGFR mutation (e.g., exon 20 insertion mutations are excluded). Enrollment of patients with mutations other than exon 19 deletion and the L858R point mutation require literature supporting sensitivity to osimertinib. T790M mutations and identified EGFR mutations that are known to confer resistance to osimertinib (for instance C797S) are allowed
* Predominantly adenocarcinoma histology. (Small cell or predominantly squamous cell or sarcomatoid/pleiomorphic histologies are excluded.)
* Progressed on osimertinib. Osimertinib must have been included in the last systemic therapy prior to trial enrollment and the patient must be considered appropriate for continuation of osimertinib at 80 mg daily per the treating investigator
* From a tumor specimen obtained following progression on osimertinib or within 4 months of study entry (as long as the specimen was obtained after osimertinib was started), subjects must have c-MET overexpressing NSCLC as assessed by a Certified Laboratory Improvement Amendments (CLIA)-certified laboratory using the VENTANA MET (SP44) RxDx assay, with intermediate or high expression, defined as either ≥ 25% and < 50% (intermediate) or ≥ 50% (high). If local results are unavailable, central testing may be performed
* Measurable disease, as per RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Able to swallow the oral study drug, has no known intolerance of study drugs or excipients, and able to comply with study requirements
* Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L
* Platelets ≥ 100 × 10^9/L
* Hemoglobin ≥ 9 g/dL
* Serum creatinine ≤1.5 X upper limit of normal (ULN) OR measured or calculated* creatinine clearance ≥ 50 mL/min (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl])

  * Creatinine clearance may be calculated using a 24 hour urine collection, by the Cockcroft-Gault formula or estimated glomerular filtration rate (eGFR) per the Modification of Diet in Renal Disease (MDRD) GFR equation
* Serum total bilirubin ≤ 1.5 X ULN OR direct bilirubin ≤ ULN
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 X ULN OR ≤ 5 X ULN for participants with liver metastases
* Albumin ≥ 3.0 g/dL
* Female participants of childbearing potential must have a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The serum test must be negative for pregnancy for the participant to be eligible. Female participants must agree to use a highly effective method of contraception from the beginning of screening until 7 months after the last dose of the telisotuzumab vedotin, or be of nonchildbearing potential.Nonchildbearing potential is defined as follows (by other than medical reasons):

  * ≥ 45 years of age and has not had menses for > 2 years, in the absence of conditions that could lead to amenorrhea (i.e., post chemotherapy),
  * Participants who have been amenorrhoeic for < 2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation, or
  * Surgical sterilization (Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation)
* Male patients having sex with a female partner of childbearing potential or a pregnant or breastfeeding partner must agree to use barrier contraception (male condom) for the duration of the treatment period until 4 months after the last dose of telisotuzumab vedotin
* Male and female participants must agree not to donate sperm or eggs, respectively starting from the first study-drug treatment, Men must not donate sperm during trial therapy and for 4 months after receiving the last dose of study medication and women must not donate eggs during trial treatment and for 7 months after receiving the last dose of study medication

Exclusion Criteria:

* Concurrent enrollment in another clinical study, unless enrolled only in the follow-up period or an observational study
* Prior c-MET targeted antibody drug conjugate with a microtubule toxin (such as monomethylauristatin E [MMAE]). Prior MET antibody without a toxin, prior MET antibody drug conjugate (ADC) with a non-microtubule, and prior MET TKI therapy are acceptable
* Any chemotherapy, immunotherapy, biologic, hormonal therapy, or investigational systemic therapy for cancer treatment in the prior 3 weeks or within 5 half-lives of the medication, whichever is shorter. Concurrent use of hormones for non-cancer-related conditions (eg, insulin for diabetes and hormone replacement therapy) is acceptable
* Thoracic radiation of ≥ 30 grey (Gy) within 6 months. Other radiation within 2 weeks with the exception: Stereotactic, palliative radiation for bone metastases is acceptable without a washout as long as no lung parenchyma was included in the radiation field
* Progressive or symptomatic brain metastases. Brain metastases that have been radiated, are asymptomatic, and on a stable or decreasing dose of steroids are allowed. Leptomeningeal disease is excluded
* Has not recovered (recovery is defined as National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events [CTCAE v 5.0] grade ≤ 1) from the acute toxicities of previous therapy, except treatment-related alopecia or laboratory abnormalities otherwise meeting the inclusion requirements stated in the inclusion criterion. Other grade 2 or less toxicities not constituting a safety risk based on the investigator's judgment are acceptable.

  * Subjects with hormone deficiencies caused by prior anticancer therapy who are asymptomatic and on a stable dose of replacement hormone are eligible for the study
* Subject must not have a history of idiopathic lung disease, drug-induced idiopathic lung disease, idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, radiation pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* Major surgical procedures or serious trauma within 4 weeks prior to cycle (C) 1 day (D) 1, or plans for major surgical procedures within 4 weeks after the first dose (as determined by the investigator). Minor local procedures (excluding central venous catheterization and port implantation) do not require a washout
* The patient has any ongoing or active infection requiring the use of parenteral anti-microbial agents. Patient with a history of HIV with an undetectable viral load and a CD4 count over 200 are eligible. Patients with a history of hepatitis B or hepatitis C, an undetectable viral load, and liver function tests (LFT) testing which meets criteria for the study are eligible
* History of another cancer within 2 years of study initiation, with the exception of fully treated cancers unlikely to affect the assessment of the study treatment safety or efficacy including early-stage breast, prostate, bladder, non-melanomatous skin, thyroid, cervical, or endometrial cancer. Additionally, subjects must not be receiving any ongoing anti-cancer therapy, including maintenance therapy, prior to randomization. Hormonal therapy is allowed provided that the participant otherwise meets trial criteria
* Participants must not be considered a poor medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to uncontrolled ventricular arrhythmia, myocardial infarction within 6 months, stroke within 6 months, clinically significant electrocardiogram (ECG) abnormalities, any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as electrolyte abnormalities, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, clinically significant liver disease, including hepatitis, current alcohol abuse, or cirrhosis, grade ≥ 2 edema or lymphedema, grade ≥ 2 ascites or pleural effusion, grade ≥ 2 neuropathy, grade ≥ 2 corneal disorder as assessed by a baseline ophthalmic exam, or any psychiatric disorder that prohibits obtaining informed consent
* Patient unwilling or unable to comply with the protocol
* Any condition that, in the opinion of the investigator or sponsor-investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  Defined as complete response or partial response per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. The ORR estimate and its associated 95% confidence interval (CI) will be calculated.
Progression free survival (PFS) | From treatment initiation to disease progression per RECIST 1.1 criteria or death, up to 2 years
  The Kaplan-Meier curve and its 95% CI will be used to infer the PFS. The median time PFS will be compared to median survival time of 4.2 months base on historic controls, using Brookmeyer-Crowley method.

SECONDARY OUTCOMES:
Duration of response | From documentation of tumor response to disease progression, up to 2 years
  The Kaplan-Meier curve and its 95% CI will be used to infer the endpoint.
Time to response | From treatment initiation until documentation of tumor response, up to 2 years
  The Kaplan-Meier curve and its 95% CI will be used to infer the endpoint.
Overall survival | From randomization to death by any cause, up to 2 years
  The Kaplan-Meier curve and its 95% CI will be used to infer the endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W Goldman, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States